CLINICAL TRIAL: NCT00960154
Title: A Prospective, Randomized, Controlled Study to Evaluate Use of the PEAK PlasmaBladeTM 4.0 in Breast Lumpectomy
Brief Title: PEAK PlasmaBlade™ 4.0 Versus Traditional Electrosurgery in Lumpectomy
Acronym: PRECISE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Termination due to acquisition of PEAK Surgical by Medtronic
Sponsor: Medtronic Surgical Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PEAK VP-00078
Record Dates: First submitted 2009-08-13; First posted 2009-08-17 (Estimated); Results first posted 2013-01-03 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Breast Cancer
Keywords: Lumpectomy; PlasmaBlade; Electrosurgery; PEAK Surgical; Medtronic Advanced Energy; Medtronic
MeSH Terms: conditions — Breast Neoplasms; Hyperthermia | interventions — Laser Therapy; Electrosurgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- PlasmaBlade (Experimental): The entirety of the lumpectomy will be performed with the PEAK PlasmaBlade, including the skin incision.
  Interventions: Device: PEAK PlasmaBlade
- SOC (Active Comparator): The SOC consists of scalpel for the skin incision and traditional electrosurgery for the entirety of the subcutaneous dissection.
  Interventions: Procedure: Traditional Electrosurgery with scalpel

INTERVENTIONS:
Device: PEAK PlasmaBlade — The entirety of the lumpectomy will be performed with the PEAK PlasmaBlade including the skin incision
  Other Names: PlasmaBlade
  Arms: PlasmaBlade
Procedure: Traditional Electrosurgery with scalpel — The skin incision will be performed using a standard scalpel; the subcutaneous dissection will be performed with traditional electrosurgery using the Cut and Coagulation modes.
  Other Names: Scalpel; Electrosurgery; SOC
  Arms: SOC

SUMMARY:
The purpose of this clinical study is to quantify the difference in thermal injury depth at the surgical margin in breast lumpectomy specimens excised with the PlasmaBlade; to subjectively assess histopathologic sample quality metrics; to examine the role that electrosurgical artifact may play in revision lumpectomy procedures; and to compare these endpoints to the standard of care (SOC) technology.

DETAILED DESCRIPTION:
Lumpectomy is a surgical procedure performed to remove a localized mass of breast tissue that is suspicious for malignancy. The purpose of lumpectomy is to minimize the amount of tissue removed from the breast to retain normal breast architecture while simultaneously removing all of the suspected cancerous tissue. Typically, a scalpel is used for the skin incision and a traditional electrosurgical device is used to cut away any cancerous tissue.

The PEAK PlasmaBlade™ uses pulsed radiofrequency (RF) energy and a highly-insulated handpiece design to enable precision cutting and coagulation at the point of application. The PlasmaBlade has received FDA clearance for use in plastic, general, and ear, nose, and throat (ENT) surgery, and has demonstrated a significantly reduced thermal injury profile in incised tissue compared to traditional electrosurgical devices. It is hypothesized that this benefit may improve the pathological analysis of excised breast lumps.

This single site study was granted Institutional Review Board (IRB) approval and conducted between June 2009 and January 2011. Potential subjects were screened against the inclusion and exclusion criteria of the study protocol and were then required to provide informed consent prior to enrollment. Following enrollment, subjects were prospectively randomized to the SOC or PEAK PlasmaBlade study groups and scheduled for lumpectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 90 years old
2. Physically healthy, stable weight
3. Requiring lumpectomy with wire localization for suspected or confirmed malignant breast disease.
4. Subject must understand the nature of the procedure and provide written informed consent prior to the procedure.
5. Subject must be willing and able to comply with all follow-up evaluations

Exclusion Criteria:

1. Age younger than 18 or greater than 90 years old
2. Infection (local or systemic)
3. Cognitive impairment or mental illness
4. Severe cardiopulmonary deficiencies
5. Unable to follow instructions or complete follow-up
6. Currently taking any medication known to affect healing
7. Currently enrolled in another investigational device or drug trial

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-07; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Naruns, MD, Principal Investigator — Midpeninsula Surgical Associates; Khoi Tran, MD, Principal Investigator — Palo Alto Medical Foundation
Locations (2):
- United States (2):
  - El Camino Surgery Center, Mountain View, California
  - Palo Alto Medical Foundation, Mountain View, California

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care (SOC): The SOC consists of scalpel for the skin incision and traditional electrosurgery for the entirety of the subcutaneous dissection.
Period: Overall Study
Arm/Group | PlasmaBlade | Standard of Care (SOC)
Started | 25 | 25
Completed | 0 | 0
Not Completed | 25 | 25
Not completed — Study termination | 25 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PlasmaBlade | Standard of Care (SOC) | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Customized [Number; unit: participants] — An integrity audit found that the data for this study could not be analyzed owing to unverifiable source documentation. The protocol-specified age range is used for this baseline measure.
  participants
    18 to 90 years | 25 | 25 | 50
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 50
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Secondary Outcome: Operative Metrics: Operative Time, Estimated Blood Loss, Skin Scarring
Time Frame: Intraoperatively and 1-2 weeks postoperatively
Population: An integrity audit found that the data for this study could not be analyzed owing to unverifiable source documentation.
Arm/Group | PlasmaBlade | Standard of Care (SOC)
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Histological Metrics: Amount of Overlying Adherent Char on Slide; Damage to Tumor Epithelium; Effect of Electrosurgical Damage on Diagnostic Quality of Lumpectomy Specimen
Description: Overall histological quality score will be a composite of the histological metrics
Time Frame: Intraoperative
Population: An integrity audit found that the data for this study could not be analyzed owing to unverifiable source documentation.
Arm/Group | PlasmaBlade | Standard of Care (SOC)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | PlasmaBlade | Standard of Care (SOC)
Serious Adverse Events (participants affected / at risk) | 1/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PlasmaBlade (N=25) | Standard of Care (SOC) (N=25)
Postoperative axillary abcess with cellulitis (Infections and infestations) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Upon Medtronic's acquisition of PEAK surgical, a study integrity audit was undertaken. Results of the audit showed that patient's rights and safety were maintained, but the source data, including baseline demographics, were unverifiable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less